CLINICAL TRIAL: NCT04248010
Title: Mechanistic Clinical Trial of Individualized tDCS for Hallucinations in Schizophrenia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Modifications in methodology had to be made that make the current registration invalid.
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Michael Avissar, Assistant Professor of Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7882
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia and Related Disorders
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Participants will receive one of the following: standard tDCS, HD-tDCS - anterior target, HD-tDCS - posterior target, or sham.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Active vs. sham will be masked; type of tDCS (standard or HD) will not be.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- standard tDCS (Active Comparator): 20 min of standard 2-electrode transcranial direct current stimulation (2 mA) at a previously reported scalp location.
  Interventions: Device: neuroConn DC-Stimulator MR
- HD-tDCS - anterior target (Active Comparator): 20 min of individualized high-density 5-electrode transcranial direct current stimulation to anterior language areas of the brain.
  Interventions: Device: Soterix MxN HD-tES
- HD-tDCS - posterior target (Active Comparator): 20 min of individualized high-density 5-electrode transcranial direct current stimulation to posterior language areas of the brain.
  Interventions: Device: Soterix MxN HD-tES
- sham tDCS (Sham Comparator): sham transcranial direct current stimulation using a brief pulse at the beginning and end of the 20 min intervention.
  Interventions: Device: neuroConn DC-Stimulator MR; Device: Soterix MxN HD-tES

INTERVENTIONS:
Device: neuroConn DC-Stimulator MR — standard tDCS, active & sham
  Arms: sham tDCS; standard tDCS
Device: Soterix MxN HD-tES — HD-tDCS, active & sham
  Arms: HD-tDCS - anterior target; HD-tDCS - posterior target; sham tDCS

SUMMARY:
This project compares standard tDCS to individualized high-definition tDCS (HD-tDCS) for treatment of auditory verbal hallucinations in schizophrenia.

DETAILED DESCRIPTION:
The large majority of patients with schizophrenia (Sz) experience auditory verbal hallucinations (AVH) as a core feature of their disorder. Treatment-resistant auditory verbal hallucinations (AVH) affect a third of patients with schizophrenia and can cause increased aggression, distress, suicide, and social dysfunction. This project will investigate the efficacy of different types of transcranial direct current stimulation (tDCS), a neurostimulation technique that passes a weak electric current through the brain, in alleviating AVH in Sz patients, and will explore hypotheses regarding brain circuits involved in AVH.

This project compares standard tDCS to individualized high-definition tDCS (HD-tDCS) for treatment of AVH. In standard tDCS, two large electrodes are positioned on the scalp above regions of the brain implicated in abnormal cortical activity associated with auditory verbal hallucinations in Sz. Due to the size of standard tDCS electrodes and the positions required to stimulate language areas, large unrelated areas of the brain are also stimulated. HD-tDCS is a novel technique that uses multiple smaller electrodes to produce a more focal electrical field (EF) than standard tDCS. The HD-tDCS used in this study modulates brain activity in a targeted area without stimulating as many unrelated areas. This targeted inhibition allows us to test hypotheses regarding different cortical regions and their roles in specific features of AVH (e.g. loudness and salience).

Participants are randomized to receive either active standard tDCS or active HD-tDCS targeting one of two language-processing areas of the brain, or a sham version of one of these stimulation types. For each participant receiving HD-tDCS, structural MRI is used to computationally model the electrical field produced in their individual brain anatomy by tDCS. These models are then used to select individualized electrode configurations and current settings to target the same language areas across subjects. The effect of stimulation on relevant brain functions is verified by measuring pre/post treatment changes in resting state functional connectivity (rsFC) within and between targeted language regions, which has been previously linked to AVH symptoms. Differences in behavioral task performance and neurophysiological abnormalities associated with AVH are also tested pre/post treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-V diagnosis of schizophrenia or schizoaffective disorder
* Capacity and willingness to provide informed consent
* Mean AHRS item score of greater or equal to 2.
* If female and not infertile, must agree to use one of the following forms of contraception for the duration of study participation: systemic hormonal treatment, an IUD which was implanted at least 2 months prior to screening, or "double-barrier" contraception. Women of child bearing potential must have a negative pregnancy test at screening
* Right handed
* Normal hearing
* Taking an antipsychotic medication at a stable dose for at least 4 weeks. All oral and depot antipsychotics are allowable.

Exclusion Criteria:

* Presence or positive history of unstable significant medical or neurological illness
* Substance use disorder (excluding nicotine) within last 90 days, or positive toxicology screen for any substance of abuse
* Pregnancy
* Participation in study of investigational medication/device within 4 weeks
* History of seizure, epilepsy in self or first-degree relatives, stroke, brain surgery, head injury with loss of consciousness >1 hour or clear cognitive sequelae, intracranial metal implants, known structural brain lesion, devices that may be affected by tDCS (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Subjects with suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the Suicidal Ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the investigator
* Frequent and persistent migraines
* Clinically significant skin disease
* Current use of medications known to lower seizure threshold (Lithium, Theophyline, Tricyclic antidepressants, Buproprion >450 mg/day and Clozapine >600 mg/day, brand name and generic methylphenidate/mixed amphetamine salts)
* History of prior clinically significant, adverse response to neurostimulation or open skin wounds that would preclude safe placement of tDCS electrodes
* Contraindication to MRI scanning, including metal implants or claustrophobia. Metal implants, pacemaker, other metal (e.g., shrapnel or surgical prostheses) or paramagnetic objects contained within the body which may present a risk to the subject or interfere with MR scan
* Medicinal patch, unless removed

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The Auditory Hallucination Rating Scale (AHRS) | 1 week
  Questionnaire-based assessment instrument for auditory verbal hallucinations, completed by study personnel.

IPD SHARING:
Plan to Share IPD: No